CLINICAL TRIAL: NCT05915286
Title: Diuretic Use in Hemodialysis Patients With Residual Renal Function: a Proof of Concept Study
Brief Title: Diuretic Use in Hemodialysis Patients With Residual Renal Function
Acronym: DIURESED
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Personnel/staffing issues.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00119451
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease on Dialysis
MeSH Terms: interventions — Furosemide; Chlorthalidone

STUDY DESIGN:
Intervention Model Description: All participants enrolled in this proof-of-concept study will be treated with the intervention (diuretic medications) in escalating doses over the study period. Each participant will act as their own control with 2 weeks of no treatment followed by the intervention for 3 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diuretic Therapy (Experimental)
  Interventions: Drug: Furosemide; Drug: Chlorthalidone

INTERVENTIONS:
Drug: Furosemide — Each participant will have a 2 week period of no diuretic use followed by 3 weeks of escalating doses: 1) initially furosemide twice daily, then (2) an increased dose of furosemide twice daily, and in the final week, (3) the addition of chlorthalidone once daily.
Drug: Chlorthalidone — Each participant will have a 2 week period of no diuretic use followed by 3 weeks of escalating doses: 1) initially furosemide twice daily, then (2) an increased dose of furosemide twice daily, and in the final week, (3) the addition of chlorthalidone once daily.

SUMMARY:
This pilot trial will evaluate the use of diuretic medications (furosemide and chlorthalidone) in participants on dialysis to see if these medications work to preserve existing kidney function, increase urine output, and reduce weight gain between dialysis treatments. Diuretics, which are sometimes called water pills, help the body to get rid of salt (sodium) and water. There are currently no guidelines for the use of diuretic medications in dialysis patients, including the type to use, or how much to use.

DETAILED DESCRIPTION:
Fluid overload, or extracellular fluid volume expansion, in patients on hemodialysis is an important predictor of mortality. It is associated with hypertension and left ventricular hypertrophy - both risk factors for cardiovascular disease. In the United States, 80% of patients receiving hemodialysis have hypertension and 40% of patients on hemodialysis die from cardiovascular disease. The pathophysiology of hypertension in these patients is multifactorial, however, combined excess fluid and sodium is a key contributor.

While ultrafiltration (removal of fluid through dialysis) is important in managing fluid overload, fluid removed by hemodialysis is a non-physiological process which imposes hemodynamic stress on the cardiovascular system in uremic patients. This system is already maladaptive as a result of decreased baroreceptor sensitivity and increased vascular stiffness, leading to higher risk of hemodynamic instability when fluid is removed from the intravascular compartment. In patients who are anuric, restriction of fluid and sodium intake and ultrafiltration are the only options for volume control. In patients who continue to produce urine, however, optimizing the amount of urine produced could improve fluid overload and decrease cardiovascular stress.

Previous studies have shown that patients on hemodialysis who have residual renal function have better volume and sodium control. Higher residual renal function and higher urine output lead to a lower interdialytic weight gain in patients receiving hemodialysis; each of these factors have been associated with lower mortality. One intervention that may increase or help maintain residual renal function and increase urine output and therefore reduce interdialytic weight gain is diuretic therapy, which promotes the excretion of sodium and water by the native kidneys. Questions remain regarding the dose-response of the drug furosemide, about the utility of adding the drug chlorthalidone, and their clinical affects.

The main objective of this study is to determine the effects of starting, and escalating doses of diuretic medications (furosemide +/- chlorthalidone) on 24-hour urine output (volume) over a five-week period in patients on hemodialysis who produce >200cc per day of urine.

Secondary objectives are:

1. To evaluate the effect of diuretic medications on residual renal function
2. To evaluate the effect of different doses of diuretics on interdialytic weight gain, ultrafiltration rates and intradialytic hypotension
3. To examine the effect of diuretics on patient reported outcomes
4. To evaluate adverse effects of different doses of diuretics
5. To measure serum furosemide levels in this patient population

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years or older), who are within their first 12 months of chronic (expected to need dialysis for at least 6 months), in-centre hemodialysis therapy, and
* Residual renal function defined as 24-hour urine volume >200cc, and
* Life expectancy of at least 6 months, and
* Participants must be able to understand the consent process and be able to sign a consent form or have a substitute decision maker who is able to understand and sign consent on their behalf. In the case of non-English speaking participants, a translator service will be used to provide study information and obtain consent.

Exclusion Criteria:

* Unable to complete baseline urine collection
* Documented allergy or adverse reaction to furosemide or chlorthalidone.
* Unable to take oral medications
* Patients expecting to change modality (peritoneal dialysis, home dialysis) or to receive a renal transplant in the next 6 weeks
* History of hypokalemia (<3.0 mmol/L), hypomagnesemia (<0.6mmol/L), or hypocalcaemia (<1.9mmol/L) in preceding 2 weeks.
* Already participating in another study and one of the studies could interfere with the other study
* Use of loop, or thiazide diuretic medications in the last week (if a patient is on chronic diuretics, they would need to be discontinued for 1 week before starting the trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour urine output | Week 1
  Change in urine output measured from 24-hour urine collection.
Change in 24-hour urine output | Week 2
  Change in urine output measured from 24-hour urine collection.
Change in 24-hour urine output | Week 3
  Change in urine output measured from 24-hour urine collection.
Change in 24-hour urine output | Week 4
  Change in urine output measured from 24-hour urine collection.
Change in 24-hour urine output | Week 5
  Change in urine output measured from 24-hour urine collection.
Change in residual renal function | Week 1
  Calculated based on weekly bloodwork (urea and creatinine levels) and 24-hour urine collection.
Change in residual renal function | Week 2
  Calculated based on weekly bloodwork (urea and creatinine levels) and 24-hour urine collection.
Change in residual renal function | Week 3
  Calculated based on weekly bloodwork (urea and creatinine levels) and 24-hour urine collection.
Change in residual renal function | Week 4
  Calculated based on weekly bloodwork (urea and creatinine levels) and 24-hour urine collection.
Change in residual renal function | Week 5
  Calculated based on weekly bloodwork (urea and creatinine levels) and 24-hour urine collection.

SECONDARY OUTCOMES:
Interdialytic weight gain | Week 1
  Patient weight measured in kilograms
Interdialytic weight gain | Week 2
  Patient weight measured in kilograms
Interdialytic weight gain | Week 3
  Patient weight measured in kilograms
Interdialytic weight gain | Week 4
  Patient weight measured in kilograms
Interdialytic weight gain | Week 5
  Patient weight measured in kilograms
Patient-reported outcomes - ESAS-r | Week 1
  Patient reported outcomes using the Edmonton Symptom Assessment System-revised (ESAS-r) questionnaire.
Patient-reported outcomes - ESAS-r | Week 2
  Patient reported outcomes using the Edmonton Symptom Assessment System-revised (ESAS-r) questionnaire.
Patient-reported outcomes - ESAS-r | Week 3
  Patient reported outcomes using the Edmonton Symptom Assessment System-revised (ESAS-r) questionnaire.
Patient-reported outcomes - ESAS-r | Week 4
  Patient reported outcomes using the Edmonton Symptom Assessment System-revised (ESAS-r) questionnaire.
Patient-reported outcomes - ESAS-r | Week 5
  Patient reported outcomes using the Edmonton Symptom Assessment System-revised (ESAS-r) questionnaire.
Patient-reported outcomes - Muscle cramps | Week 1
  Patient reported outcomes using a muscle cramps question.
Patient-reported outcomes - Muscle cramps | Week 2
  Patient reported outcomes using a muscle cramps question.
Patient-reported outcomes - Muscle cramps | Week 3
  Patient reported outcomes using a muscle cramps question.
Patient-reported outcomes - Muscle cramps | Week 4
  Patient reported outcomes using a muscle cramps question.
Patient-reported outcomes - Muscle cramps | Week 5
  Patient reported outcomes using a muscle cramps question.
Adverse effects | Week 1
  Adverse effects based on symptoms and weekly bloodwork.
Adverse effects | Week 2
  Adverse effects based on symptoms and weekly bloodwork.
Adverse effects | Week 3
  Adverse effects based on symptoms and weekly bloodwork.
Adverse effects | Week 4
  Adverse effects based on symptoms and weekly bloodwork.
Adverse effects | Week 5
  Adverse effects based on symptoms and weekly bloodwork.
Urine furosemide levels | Week 3
  Urine furosemide levels from weekly urine samples
Urine furosemide levels | Week 4
  Urine furosemide levels from weekly urine samples
Urine furosemide levels | Week 5
  Urine furosemide levels from weekly urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Branko Braam, MD/Ph.D., Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No